CLINICAL TRIAL: NCT03934788
Title: A Prospective Randomized Controlled Study to Evaluate the Clinical Performance of OxySoft Silicone Hydrogel Soft Contact Lens
Brief Title: the Clinical Performance of the Oxysoft Daily Disposable Silicone Hydrogel Soft Contact Lens
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visco Vision Inc. (Industry)
Collaborators: Jens Medical Consulting Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 1060510M
Record Dates: First submitted 2019-04-29; First posted 2019-05-02 (Actual); Last update posted 2019-05-02 (Actual); Status verified 2019-04

CONDITIONS: Myopia
Keywords: contact lens material; silicon hydrogel
MeSH Terms: conditions — Myopia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Oxysoft (Experimental): olifilcon C, daily disposable soft contact lens, 1 month
  Interventions: Device: oxysoft (olifilcon C)
- SiHy (Active Comparator): olifilcon B, dialy disposable soft contact lens, 1 month
  Interventions: Device: Si-Hy (olifilcon B)

INTERVENTIONS:
Device: oxysoft (olifilcon C) — subjects meet certain criteria will be administered randomly oxysoft on both eye for one month on daily wear single use modality.
  Arms: Oxysoft
Device: Si-Hy (olifilcon B) — subjects meet certain criteria will be administered randomly Si-Hy on both eye for one month on daily wear single use modality.
  Arms: SiHy

SUMMARY:
The objective of this study is to demonstrate that the OxySoft silicone hydrogel soft contact lens could be prescribed as a supportive care for myopes.

DETAILED DESCRIPTION:
This is a double blind randomized control study to evaluate a daily disposable contact lens. It is planned to have 30 evaluable subjects at least divided evenly among 3 independent PIs. Each PI will enroll 12 subjects at least. The ration of evaluable test subjects to control subjects will be 2 to 1. The study lens will be dispensed randomly to subjects who have normal ocular health and conform to a set of criteria. It is necessary to wear the lens 8 hours a day and 5 days a week at least and follow up for one month (30 days). Data will be collected at baseline, 1 week, 2 week and 4 week of daily disposable modality including Adverse Reactions, Slit-lamp findings and Symptoms, Problems, and Complaints, vision acuity, keratometry change and reason for discontinuation.

ELIGIBILITY:
Inclusion Criteria:

* Subject should have normal eye and use no ocular medications
* VA correctable to 0.1 LogMAR or better, with spherical lenses ranging in power from -1.00 to -10.00 D myopia, astigmatism =< 2.00 D
* Willing to comply with all study procedures and be available for the duration of the study.
* Provide signed and dated informed consent form.

Exclusion Criteria:

* Subjects have history of allergies that would contraindicate "normal" contact lens wear.
* Subjects have other active ocular or systemic disease such as, but not limited to: anterior uveitis (past or present), glaucoma, Sjögren's syndrome, lupus erythematosus, sclerodermas, keratoconus or type II diabetes, slip lamp findings greater than grade I (such as cornea or interstitial edema).
* Subjects have medications that would contraindicate contact lens wear.
* The presence of clinically significant (grade 3 or 4) anterior segment abnormalities; inflammations such as iritis; or any infection of the eye, lids, or associated structures.
* A known history of corneal hypoesthesia (reduced corneal sensitivity), corneal ulcer, corneal infiltrates or fungal infections.
* A history of papillary conjunctivitis that has interfered with contact lens wear.
* Any active participation in another clinical trial within 30 days prior to this study.
* Have had any cornea surgery.
* Currently pregnant (to the best of the subject's knowledge), is lactating or is planning a pregnancy within the next 1 month.
* Monocular or monovision fits
* Alcoholic or Drug Abused.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-09-26 (Actual); Primary Completion 2018-11-29 (Actual); Study Completion 2018-11-29 (Actual)

PRIMARY OUTCOMES:
Log MAR visual acuities | 1 month
  The primary efficacy will be Log MAR visual acuities (VA) of 0.1 or better.

SECONDARY OUTCOMES:
slit lamp findings | 1 month
  Any slit lamp findings > grade 2 [ Time Frame: over all follow-up visits for the 1 month ] slit lamp findings on all dispensed eyes over all follow-up visits. Measured on a scale of 0-4 with 0=no findings and 4=sever findings.

CONTACTS AND LOCATIONS:
Overall Officials: Huey Chuan Cheng, MD MSc, Principal Investigator — Mackay Memorial Hospital
Locations (3):
- Taiwan (3):
  - Taipei TzuChi Hopsital, Buddhist Tzu Chi Medical Foundation, New Taipei City
  - Tri-Service General Hospital_Tingjhou, Taipei
  - MayKay Memorial Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No